CLINICAL TRIAL: NCT01834066
Title: Safety and Efficacy of Bone Marrow Autologous Cells in Muscular Dystrophy. It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Study Safety and Efficacy of Bone Marrow Derived Autologous Cells for the Treatment of Muscular Dystrophy.
Acronym: mdp
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, C0- Investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00101
Record Dates: First submitted 2013-02-26; First posted 2013-04-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Muscular Dystrophy; Duchenne Muscular Dystrophy,
Keywords: muscular Dystrophy stem cell
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- STEM CELL (Other): Intra thecal transplantation of autologous Stem Cell MNCs
  Interventions: Biological: Stem Cell

INTERVENTIONS:
Biological: Stem Cell — Intralesional transfer of Autologous Stem cell (MNCs) per dose. 6 doses in 3 months
  Other Names: Intravenous transfer of Autologous Stem Cell ( MNCs )

SUMMARY:
This Study is single arm, single centre trial to check the safety and efficacy of Bone Marrow derived autologous cell(100 million per dose) for the patient with Duchenne Muscular Dystrophy.

DETAILED DESCRIPTION:
Muscular dystrophy is a group of inherited disorders that involve muscle weakness and loss of muscle tissue, which get worse over time. Duchenne muscular dystrophy is caused by a defective gene for dystrophin (a protein in the muscles). However, it often occurs in people without a known family history of the condition. slowly progress diseases.it causes Muscle weaknesses, Difficulty with motor skills ,Progressive difficulty walking.Breathing difficulties and heart disease,Frequent falls,weak limbs,lose motor Function.Begins in the legs and pelvis, but also occurs less severely in the arms, neck, and other areas of the body.Trouble getting up from a lying position or climbing stairs.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Diagnose of Duchenne Muscular Dystrophy.
* Aged in between 6 to 25 Years.
* Willingness to undergo Bone Marrow derived Autologous cell Therapy.
* Ability to comprehend the explained protocol and thereafter give an informed consent as well as sign the required Informed Consent form(ICF) for the study.
* Ability and willingness to regular visit to hospital for protocol procedures and follow up

Exclusion Criteria:

* Patient who is not Diagnose of Duchenne Muscular Dystrophy.
* Patient with History of Immunodeficiency HIV+,Hepatitis B ,HBV and TPPA+,Tumor Markers+
* History of Life threatening allergic or immune -Mediated Reaction.
* the site of bone marrow aspiration potentially limiting Procedure.
* Alcohol and drug abuse / dependence.
* Patients with History of Hypertension and Hypersensitive.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Significant Improvement in Muscle strength by using Kinetics Muscle testing or by using MMT( manual muscle test }score | 6 Months

SECONDARY OUTCOMES:
-Improvement of daily living scale and baseline in EMG(electromyography) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, MS ORTHO, Principal Investigator — CHAITANYA HOSPITAL
Locations (1):
- Chaitnany Hospital, Pune, Maharashtra, India